CLINICAL TRIAL: NCT00693888
Title: Lighthouse Project on Dementia, Ulm, Germany - Improvement of Advice and Diagnostics for People Suffering From Dementia After the Classification of Their Level of Care (ULTDEM Study).
Brief Title: Lighthouse Project on Dementia, Ulm, Germany
Acronym: ULTDEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government); Geriatric Center Ulm (Unknown); Robert Bosch Medical Center (Other)
Responsible Party: Thorsten Nikolaus, M.D. professor, Geriatric Center Ulm (GZU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LTDemenz-44-052
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2009-03

CONDITIONS: Dementia
Keywords: dementia; system of care; level of care; interventional study; evaluation; dementia diagnostic; Evaluation of the care study
MeSH Terms: conditions — Dementia | interventions — Counseling; Jurisprudence; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interventional group (Experimental): individual comprehensive primary advice (e.g. medical and social aspects, care, support at home, residential advice, legal aspects, demonstration of help and support for the relatives)
  Interventions: Behavioral: advice (e.g. medical and social aspects, care, support at home, residential advice, legal aspects, demonstration of help and support for the relatives)
- Control group (No Intervention): only informative flyer, no further advice in any direction

INTERVENTIONS:
Behavioral: advice (e.g. medical and social aspects, care, support at home, residential advice, legal aspects, demonstration of help and support for the relatives) — initial comprehensive assessment, stratified (city, suburbs) randomization into two groups: interventional group: individual comprehensive primary advice (medical and social aspects, care, support at home, residential advice, legal aspects, demonstration of help and support for the relatives), control group: standard support, observation over a period of 6 months, possibility of completing the diagnostic after final assessment
  Arms: interventional group

SUMMARY:
The Geriatric Center Ulm scientifically supported a three-year pilot study (ProjektDEMENZ Ulm), in which numerous findings on the system of care regarding people suffering from dementia and their relatives were determined.

One of the most important conclusions is the significant lack of information on the well-functioning network of the care system in Ulm. The full potential of the network is not being exploited.

The situation in the Alb-Donau-Kreis - the area surrounding Ulm - is very similar.

The investigators' aim is to improve the utilization of the system of care for those suffering from dementia in Ulm/Alb-Donau-Kreis by using a newly designed advisory approach (Lighthouse Project on Dementia, Ulm, ULTDEM study).

The purpose of the study is to prove the effectiveness of this procedure by using a prospective, open, randomized, controlled, interventional study.

After the randomization, the interventional group is given comprehensive, individual advice about available treatment possibilities for people suffering from dementia.

In addition, they have the opportunity to re-evaluate their present diagnostic procedure.

The participants of the control group receive the standard treatment. Inclusion criterion is the application of a care level ( level 0 or 1). Recruitment will take one year. A final assessment will be taken every six months.

ELIGIBILITY:
Inclusion Criteria:

* dementia (MMSE < 24)
* signing up for classification of care level (0 or 1)
* community dwelling elderly (older than 60 years)
* member of certain health insurance provider (AOK, Barmer, DAK)
* residents of Ulm / Alb-Donau-Kreis

Exclusion Criteria:

* result from the inclusion criteria
* cancer
* consuming disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-02 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life | six months

SECONDARY OUTCOMES:
health economical effects, progress of disease, level of evidence based on diagnosis, institutionalization, hospitalization, using support possibilities, use of drugs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Nikolaus, M.D., professor, Principal Investigator — Geriatric Center Ulm / Alb-Donau (GZU)
Locations (1):
- Geriatric Center Ulm (GZU), Bethesda Geriatrische Klinik Ulm, Ulm, Baden-Wurttemberg, Germany